CLINICAL TRIAL: NCT07121374
Title: NEoadjuvant Chemotherapy and Immunotherapy for a Selected Group of Inoperable Pleural Mesothelioma Patients (NECIM): a Feasibility Study
Acronym: NECIM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: University Hospital, Ghent (Other); Kom Op Tegen Kanker (Other)
Responsible Party: Principal Investigator, Jeroen Hendriks, PhD & MD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2387; 2023-504302-11-02 (EU CTIS Number)
Record Dates: First submitted 2025-07-25; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pleural Epithelioid Mesothelioma; Mesothelioma; Pleura; Neoadjuvant Chemoimmunotherapy
Keywords: NECIM
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cerebral Decortication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): systemic treatment and surgery
  Interventions: Drug: Neoadjuvant chemo-immunotherapy; Procedure: Extended pleurectomy/decortication in case of reaching operability

INTERVENTIONS:
Drug: Neoadjuvant chemo-immunotherapy — Neoadjuvant chemotherapy (2 cycles of cisplatin OR carboplatin accord healthcare- investigator's choice - PLUS pemetrexed fresenius AND immunotherapy (2 cycles of Opdivo PLUS 1 cycle of Yervoy for inoperable T2-T3 TNM 9 patients with PM
Procedure: Extended pleurectomy/decortication in case of reaching operability — After the systemic treatment the surgery will follow if patient is operable.

SUMMARY:
The goal of this clinical trial is to evaluate whether a combination of chemotherapy and immunotherapy can make surgery possible in adults with inoperable pleural mesothelioma (a type of cancer affecting the lung lining). The main questions it aims to answer are:

Can two cycles of neoadjuvant chemotherapy and dual immunotherapy, followed by surgery, be completed safely and effectively?

Does this treatment allow previously inoperable patients to become eligible for surgery and improve survival outcomes?

Participants will:

Receive two cycles of chemotherapy (cisplatin or carboplatin and pemetrexed)

Receive dual immunotherapy (nivolumab and ipilimumab)

Undergo evaluation by a multidisciplinary team to determine if surgery is possible

If operable, undergo extended pleurectomy/decortication surgery

Be followed for one year to assess side effects, quality of life, and survival

ELIGIBILITY:
Inclusion Criteria:

* Capable of written informed consent and adherence to study procedures
* Pathologically confirmed PM (epithelioid), cT2-3 N0-1 M0 according to UICC TNM 9 and considered inoperable by the Multidisciplinary Tumor Board of UZA/UZG at the start of the trail. They only enter the second surgical stage when becoming operable after neoadjuvant therapy
* Aged 18 years or older
* World Health Organization (WHO) Performance Status 0-1
* Fit for systemic chemotherapy, immunotherapy and surgery according to good clinical practice
* No pregnancy allowed: women of childbearing potential have to take adequate contraception to avoid pregnancy; men need to take adequate contraception (usage of a condom) to avoid pregnancy in female partners

Exclusion Criteria:

* Operable PM patients according to TNM 9 criteria (T1) or inoperable PM patients who will not have a chance to become operable after neoadjuvant treatment according to TNM 9 criteria (some T3, all T4, N2-3, M1)
* Contralateral mediastinal (N2) or distant metastatic disease (evaluated by PET and chest CT)
* Patients unfit for systemic chemotherapy, immunotherapy or intrathoracic surgery. Patients with an active autoimmune disease or who have had prior splenectomy, an active/acute infection requiring antibiotics, a chronic infection (e.g. HIV, hepatitis B or C) or have a serious cardiac disease are unfit for systemic therapy because their immune system is not properly functioning
* Hypersensitivity or contraindications to the active substance or to any of the excipients of the medications (platinum salts, pemetrexed, ipilimumab, nivolumab) used in this study
* Concurrent active malignancy other than basal cell carcinoma of the skin or in situ carcinoma of the cervix including brain metastases
* Prior treatment with chemotherapy, immunotherapy, surgery (except for diagnostic thoracoscopy) or thoracic RT (including prophylactic tract irradiation)
* Patients with significantly altered mental status or with psychological, familial, sociological or geographical conditions potential hampering compliance with the study as decided by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
To assess the percentage of successful completion of a neoadjuvant double chemotherapy / double immunotherapy regimen followed by surgery in a selected group of T2-T3 (according to TNM 9) patients with pleural mesothelioma. | The primary end point will be measured on week 17 +/-2 weeks
  The primary endpoint is the rate of success, which is defined as a composite endpoint of feasibility, efficacy and safety consisting of:
  Feasibility is defined at week 17 +/- 2 weeks after start of treatment and involves the successful completion of 2 cycles of neoadjuvant immunotherapy and chemotherapy, being selected as operable thereafter, and having extended pleurectomy/decortication (P/D).
  AND Efficacy is defined as being alive and without signs of progressive disease at week 17 +/- 2 weeks after start of treatment AND Safety is defined as absence of grade 3-4 residual toxicity from systemic treatment and complete resolution of major complications (grade III - V) after surgery according to the Ottawa Thoracic Surgery Morbidity and Mortality Classification at week 17 +/- 2 weeks after start of treatment Patients who are still inoperable after successful completion of 2 cycles of neoadjuvant immunotherapy and chemotherapy are considered failure for the primary endp

SECONDARY OUTCOMES:
Toxicity of the neoadjuvant double chemotherapy / double immunotherapy regimen and surgery. | The End of Treatment will be at 17 weeks
  Toxicity, assessed by CTC-AE scores. Chemotherapy and immunotherapy-related toxicity assessed using the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. At the end of Treatment on week 17 ± 2 weeks). The CTCAE Grade (1-5); higher scores indicate more severe adverse events.
Toxicity of the neoadjuvant double chemotherapy / double immunotherapy regimen and surgery. | The End of Treatment will be at 17 weeks
  Toxicity, assessed by the Ottawa scores for surgery.
  Postoperative surgical complications are assessed using the Ottawa Thoracic Morbidity and Mortality Classification. At End of Treatment on week 17 ± 2 weeks, including postoperative period. The Ottawa classification Grade (I-V); higher grades indicate more severe complications.
Efficay of neoadjuvant double chemotherapy / double immunotherapy regimen in inoperable T2-3 PM patients. | operability will be evaluated after systemic treatment on week 7-9.
  Efficacy, assessed by the percentage of T2 and T3 PM patients becoming operable after double neoadjuvant chemotherapy and immunotherapy which is defined by the radiology department using the TNM 9 criteria.
Quality of life during the neoadjuvant double chemotherapy / double immunotherapy regimen and surgery. | at week 17
  Quality of life, assessed by the EQ-5D-5L score. The EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L), a standardized instrument for measuring health-related quality of life. The EQ-5D-5L consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 5 response levels. In addition, it includes a visual analogue scale (EQ-VAS) for self-rated health.
  Time Frame: At baseline, Day 1 of each treatment cycle, pre-surgery, End of Treatment (Week 17 ± 2 weeks), and follow-up visits at Weeks 13, 26, 39, and 52 after EoT.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium